CLINICAL TRIAL: NCT02320539
Title: MicroRNA Diagnostics in Subarachnoid Hemorrhage 2
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Søren Bache, MD, MD, Rigshospitalet, Denmark
Other Study IDs: H-6-2014-073
Record Dates: First submitted 2014-10-28; First posted 2014-12-19 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Subarachnoid Hemorrhage; Delayed Cerebral Ischemia; Acute Lung Injury; Cardiac Dysfunction; Systemic Inflammatory Response Syndrome
Keywords: MicroRNA; Cerebrospinal fluid
MeSH Terms: conditions — Subarachnoid Hemorrhage; Acute Lung Injury; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — MicroRNA profiles from blood and cerebrospinal fluid are investigated.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- SAH with DCI: After 21 days from ictus the patients with subarachnoid hemorrhage are stratified to group 1 or 2 depending on their development of delayed cerebral ischemia.
- SAH without DCI: After 21 days from ictus the patients with subarachnoid hemorrhage are stratified to group 1 or 2 depending on their development of delayed cerebral ischemia.
- SAH good grade: SAH without external ventricular drainage
- Healthy controls: Blood sample in healthy donors registered in the National Donor Registry.

SUMMARY:
The purpose of this study is to validate results from a related trial (NCT01791257) and to compare the profile of microRNA in blood from patients suffering subarachnoid hemorrhage with and without systemic complications.

DETAILED DESCRIPTION:
In this study of patients suffering an aneurysmal subarachnoid hemorrhage (SAH) we would like to validate former results from CSF studies through microRNA profiling investigate the pathophysiological mechanisms that lead to systemic complications such as cardiac dysfunction, acute lung injury (ALI) and systemic inflammatory response syndrome(SIRS).

We will accomplish this through analyzing the profile of microRNA expression in blood and cerebrospinal fluid from SAH patients.

Validation:

As in our earlier study we wish to compare the expression of 20 specific microRNA between 12 patients developing DCI (group 1) and 12 patients without DCI (group 2) in cerebrospinal fluid drawn on day 5 after ictus. In addition, some of the patients will have established invasive neuromonitoring including microdialysis in which we will study changes of certain microRNAs.

DCI as defined by Vergouwen et al in Stroke 2010;41(10):2391-2395:

"The occurrence of focal neurological impairment (such as hemiparesis, aphasia, apraxia, hemianopia, or neglect), or a decrease of at least 2 points on the Glasgow Coma Scale (either on the total score or on one of its individual components [eye, motor on either side, verbal]). This should last for at least 1 hour, is not apparent immediately after aneurysm occlusion, and cannot be attributed to other causes by means of clinical assessment, CT or MRI scanning of the brain, and appropriate laboratory studies."

Systemic complications:

Furthermore, we wish to compare the expression of 754 specific microRNA in blood drawn on day 3 after ictus between patients with ALI (as described Kahn et al, Crit Care Med. 2006; 34: 196-202) and patients without ALI. Of at least 36 patients expected to be included 12 should statistically develop ALI according to the referred definition.

Additionally, we wish to compare the expression of 754 specific microRNA between 12 patients developing DCI (group 1) and 12 patients without DCI (group 2) in blood drawn on day 3 after ictus.

Moreover, we wish to compare the expression of 754 specific microRNA in blood between 36 patients (group 1-3) to that of healthy controls. The specific microRNAs of interest in which the expression in blood between patients with systemic complication are analyzed daily to investigate the dynamic changes in expression and compared to the clinical course.

ELIGIBILITY:
Inclusion Criteria Group 1-3:

* Uncertainty < 24 times on time of ictus

Inclusion Criteria Group 1-2:

* Patients admitted to Neurointensive Department in Rigshospitalet with aneurysmal SAH treated with external ventricular drain.

Inclusion Criteria Group 3:

* Patients admitted to Neurointensive Department in Rigshospitalet with aneurysmal SAH treated without external ventricular drain.

Exclusion Criteria Group 1-3:

* Transfer to other hospital within 5 days of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1-2: Patients admitted to Neurointensive Department in Rigshospitalet with SAH treated with external ventricular drain.
  Group 3: Patients admitted to Neurointensive Department in Rigshospitalet with SAH treated without external ventricular drain.
  Group 4: Healthy blood donors
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Delayed Cerebral Ischemia | 21 days
  Delayed Cerebral Ischemia as defined by Vergouwen et al[1]. In our earlier study we found the clinical condition DCI somehow subjective which is why we added the following two primary outcome measures.
  Comparing microRNA profiles between groups with or without.
Delayed Cerebral Ischemia and Cerebral infarction | 21 days
  as defined by Vergouwen et al [1].
  Comparing microRNA profiles between groups with or without.
Delayed Cerebral infarction | 21 days
  as defined by Vergouwen et al [1].
  Comparing microRNA profiles between groups with or without.

SECONDARY OUTCOMES:
Acute Lung Injury | 21 days
  as defined by Kahn et al[2].
  Comparing microRNA profiles between groups with or without
Cardiac Dysfunction | 21 days
  Evaluated by transthoracic echocardiography
  Comparing microRNA profiles between groups with or without
Systemic Inflammatory Response Syndrome | 21 days
  Evaluated through daily vital signs and biochemistry
  Comparing microRNA profiles between groups with or without
Early Brain Injury | Clinical evaluation 24-72 hours after ictus. (Wake-up call if sedated)
  Early Brain injury = GCS 3-12 and/or paresis (degree 4) of at least one extremity or aphasia No Early Brain injury = GCS 13-15 and no or only small and mild focal deficit
  Comparing microRNA profiles between groups with or without

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Møller, Prof, Study Director — Neurointensive Care Unit, The Neuroscience Center, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark, Denmark

REFERENCES:
- [Derived] Matzen JS, Krogh CL, Forman JL, Garred P, Moller K, Bache S. Lectin complement pathway initiators after subarachnoid hemorrhage - an observational study. J Neuroinflammation. 2020 Nov 12;17(1):338. doi: 10.1186/s12974-020-01979-y. PMID 33183322
- See also: [1] Vergouwen et al in Stroke 2010;41(10):2391-2395. — http://www.ncbi.nlm.nih.gov/pubmed/?term=20798370
- See also: [2] Kahn et al, Crit Care Med, Vol. 34, No.1 2006 — http://www.ncbi.nlm.nih.gov/pubmed/16374174